CLINICAL TRIAL: NCT00161980
Title: A Randomized and Controlled Clinical Study to Evaluate the Efficacy and Safety of Fibrin Sealant VH S/D (FS VH S/D) in Reduction of Lymphatic Leakage by Sealing Axillary Lymph Node Dissection Sites
Brief Title: Efficacy and Safety of Fibrin Sealant Vapor Heated Solvent/Detergent Treated (FS VH S/D) for Reduction of Lymphatic Leakage by Sealing Axillary Lymph Node Dissection Sites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550002
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-10-23 (Estimated); Status verified 2006-10

CONDITIONS: Breast Cancer; Lumpectomy; Mastectomy Plus Axillary Lymph Node Dissection; Lymphatic Leakage
Keywords: Axillary wound; Seroma; Fistulae
MeSH Terms: conditions — Breast Neoplasms; Seroma | interventions — Surgical Procedures, Operative

INTERVENTIONS:
Drug: Fibrin Sealant VH S/D
Procedure: Surgical intervention alone without Fibrin Sealant VH S/D application

SUMMARY:
This study will monitor the safety of FS VH S/D and will evaluate whether FS VH S/D is superior to conventional surgical procedures in the reduction of lymphatic leakage by sealing the axillary lymphatics in subjects undergoing lumpectomy and level I and II axillary lymph node dissection with two separate incisions.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained from the subject prior to FS VH S/D administration
* Female subjects >= 19 years of age
* Subjects with breast cancer scheduled to undergo lumpectomy of the breast and level I and II axillary lymphadenectomy with two separate incisions

Exclusion Criteria:

* Subjects with known hypersensitivity to aprotinin or other components of the product
* Subjects with immunodeficiency
* Subjects with increased red cell production (e.g., in hemolytic anemia)
* Subjects with coagulation disorders shown by exceeding the normal range of any of following: prothrombin time (PT), Quick, activated partial thromboplastin time (aPTT), fibrinogen level, or thrombocytes.
* Subjects having previously had axillary surgery
* Subjects having undergone irradiation therapy to the axillary tissue
* Subjects having ever received chemotherapy before the surgery

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Berger, MD, Principal Investigator — General Hospital / University Hospital Vienna, Austria; Diethelm Wallwiener, MD, Principal Investigator — University of Tübingen, Germany
Locations (8):
- Austria (2):
  - Landeskrankenhaus St. Pölten, Sankt Pölten, Lower Austria
  - Allgemeines Krankenhaus der Stadt Wien, University Clinic for Gynecology, Vienna
- Centre Régional de Lutte Contre le Cancer, Centre Eugène Marquis, Rennes, France
- Germany (3):
  - Ludwig-Maximilians-Universität, Munich
  - Universitätsklinikum Tübingen, Frauenklinik, Tübingen
  - Universitätsklinikum - Frauenklinik, Würzburg
- Italy (2):
  - S. Luigi - S. Curro, Presidi Ospedalieri Unificati, Catania
  - Istituto Nationale per la Ricerca sul Cancro, Genova